CLINICAL TRIAL: NCT02445755
Title: Transcutaneous Bilirubinometry in Neonates With the Bilicare System
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vinod K. Bhutani, MD, Stanford University
Other Study IDs: 30820; NCT02372045 (obsolete NCT alias)
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-05

CONDITIONS: Transcutaneous Bilirubinometry
Keywords: Neonates; Bilicare System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to test the performance of a new transcutaneous ("measured through skin") bilirubin device (BiliCare™) to measure bilirubin levels. The investigators plan to evaluate the clinical performance of this device as a point of care test. If the investigators can validate the BiliCare™ with bilirubin from your baby's blood they could verify a non-invasive alternative for measuring bilirubin.

ELIGIBILITY:
Inclusion Criteria:

1. Parental informed consent
2. Male and female newborns with a GA ≥ 35 wks
3. Enrollment at age > 6 hrs until neonatal discharge
4. Pre-phototherapy

Exclusion Criteria:

1. Infants requiring respiratory assistance (such as mechanical ventilation)
2. Severe or life-threatening congenital anomalies
3. Hematomas at the point of measurement on both ears
4. Neonates undergone blood transfusion

Min Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 100 total participants will be enrolled by the study. Since the goal of the study is to ASSAY SAMPLE FROM BABIES WITH DIVERSE BILIRUBIN LEVELS, the study participants will be moderate premature and mature infants. In particular, the target population will be moderate premature infants at >35 weeks postmenstrual age (PMA) and of term PMA.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Late Preterm and Term Newborns: The study population will consist of term and late preterm newborns (infants >=35 weeks gestational age)
Period: Overall Study
Arm/Group | Late Preterm and Term Newborns
Started | 113 (Neonates will be tested with 3 transcutaneous (TcB) devices +/-30 minutes of routine bilirubin labs)
Completed | 100
Not Completed | 13
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 6
Not completed — Screen Failure | 5

BASELINE CHARACTERISTICS:
Arm/Group | Late Preterm and Term Newborns
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Gestational Age (GA) in weeks
  Weeks | 38 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 1
  White | 41
  More than one race | 0
  Unknown or Not Reported | 36

OUTCOME MEASURES:

1. Primary Outcome: In This Study, the Investigators Plan to Test the Performance of a Novel Transcutaneous Device (BiliCareTM) to Screen for Bilirubin Levels at Postnatal Age of 12 to 48 Hours.
Time Frame: 12 to 48 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- BiliCare TcB: The study population will consist of term and late preterm newborns (infants >=35 weeks gestational age) measured with the BiliCare TcB device
- BiliCare TcB With Infection Control Tip: The study population will consist of term and late preterm newborns (infants >=35 weeks gestational age) measured with the BiliCare TcB device with infection control tip.
- JM103 TcB: The study population will consist of term and late preterm newborns (infants >=35 weeks gestational age) measured with the JM103 TcB device
- Total Serum Bilirubin (TSB): The study population will consist of term and late preterm newborns (infants >=35 weeks gestational age) measured routinely for total serum bilirubin by diazo method.
Arm/Group | BiliCare TcB | BiliCare TcB With Infection Control Tip | JM103 TcB | Total Serum Bilirubin (TSB)
Number analyzed (Participants) | 100 | 100 | 97 | 100
mg/dL | 7.5 (2.7) | 7.6 (2.9) | 6.1 (3.0) | 6.4 (3.2)

ADVERSE EVENTS:
Arm/Group | Late Preterm and Term Newborns
Serious Adverse Events (participants affected / at risk) | 0/113
Other Adverse Events (participants affected / at risk) | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No